CLINICAL TRIAL: NCT03156777
Title: A Single Center Observational Study to Evaluate the Application Value of Circulating Tumor Cell Detection for Advanced Gastric Cancer Patients in Prediction of the Prognosis and Evaluation of the Outcome of Adjuvant Chemotherapy
Brief Title: Application Value of CTCs Detection for Advanced Gastric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-16-038
Record Dates: First submitted 2016-11-30; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2016-11

CONDITIONS: Circulating Tumor Cells; Gastric Cancer
Keywords: Gastric cancer; Circulating tumor cells; Prognosis
MeSH Terms: conditions — Neoplastic Cells, Circulating; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluating the application value of a new circulating tumor cell detection method for advanced gastric cancer patients in prediction of the prognosis and early evaluation of the result of postoperation adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment must meet all of the following criteria:

1. Provide signed informed consent. The subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign informed consent, approved by the Independent Ethic Committee (IEC)/Institutional Review Board (IRB) prior to the initiation of any study-specific procedures
2. Men or women aged >= 18 years and <=75 years.
3. Eastern Cooperative Oncology Group Performance Status (ECOG) <= 2.
4. Histologically confirmed adenocarcinoma of the stomach, gastroesophageal junction.
5. Metastatic disease or locally advanced disease not amenable to curative surgery.
6. Radiographically assessable, non-measurable disease or measurable disease as per RECIST criteria.
7. Life expectancy of at least 12 weeks with tumor and at least 5 years without tumor from the time of enrollment.
8. No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
9. No prior chemotherapy for advanced disease. -

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Gastric carcinoid, sarcomas, or squamous cell cancer.
2. Pregnant or lactating females.
3. Significant neurological or psychiatric disorders (psychotic disorders, dementia or seizures) that would prohibit the understanding and giving of informed consent.
4. Active Hepatitis B or C or history of an HIV infection.
5. Active uncontrolled infection. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced gastric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of circulating tumor cell (CTC) | Up to 2 years from start of study
  Number of the circulating tumor cell in peripheral blood from advanced gastric cancer patients undergoing D2 radical resection followed by first-line chemotherapy

SECONDARY OUTCOMES:
Profile and Portion of circulating tumor cell (CTC) | Up to 2 years from start of study
  Profile and Portion of the circulating tumor cell in peripheral blood from advanced gastric cancer patients undergoing D2 radical resection followed by first-line chemotherapy. There are three type of CTCs: epithelial type CTC，mesenchymal type CTC and mixed type CTC. The portion of different type of CTC were calculated, for example: the portion of epithelia type CTC number to total CTCs,etc.
Progression-free survival | Up to 3 years from start of the study
  Survival duration since radical resection to clinical finding of relapse disease.
Overall survival | Up to 5 years from start of the study
  Survival duration since radical resection to patient die.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, M.D. & Ph.D., Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Yinbing Liu, M.D. & Ph.D., Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided